CLINICAL TRIAL: NCT00689559
Title: A Single-Centre, Double-Blind, Randomised, Parallel Group Study of Repeated Oral Doses of AZD3480/Placebo and a Single Dose of Aripiprazole to Evaluate the Pharmacokinetic Interaction Between AZD3480 and Aripiprazole in Healthy Subjects (Phase I)
Brief Title: Drug Interaction Study Between AZD3480 and Aripiprazole in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Hans-Göran Hårdemark, MD, PhD, Medical Science Director, AstraZeneca R&D Södertälje
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: D3691C00001; EudraCt nr 2008-000310-74
Record Dates: First submitted 2008-05-29; First posted 2008-06-03 (Estimated); Last update posted 2009-07-02 (Estimated); Status verified 2009-06

CONDITIONS: Alzheimer's Disease
Keywords: Alzheimer's disease; AZD3480; Aripiprazole
MeSH Terms: conditions — Alzheimer Disease | interventions — ispronicline; Aripiprazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): AZD3480 + Aripiprazole
  Interventions: Drug: AZD3480; Drug: Aripiprazole
- 2 (Experimental): Placebo + Aripiprazole
  Interventions: Drug: Placebo; Drug: Aripiprazole

INTERVENTIONS:
Drug: AZD3480 — AZD3480 capsules qd, oral, 22 days
  Arms: 1
Drug: Placebo — Placebo qd, 12 days
  Arms: 2
Drug: Aripiprazole — single dose on day 5
  Other Names: Abilify

SUMMARY:
The purpose of the study is to evaluate if AZD3480 and warfarin interact with each other or not, i.e. show the same or altered plasma concentration profiles when co-administered compared to administered alone.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed written informed consent
* Clinically normal physical findings and laboratory values

Exclusion Criteria:

* Clinically significant illness or clinically relevant trauma within three weeks before the first dose
* History of clinically significant disease
* Use of prescribed medication during the 2 weeks before administration of the first dose of investigational product

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Estimated)
Dates: Start 2008-03; Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
PK variables | Frequent sampling occasions during

SECONDARY OUTCOMES:
Safety variables (adverse events, blood pressure, pulse, safety lab) | During the whole treatment period

CONTACTS AND LOCATIONS:
Overall Officials: Lennart Jeppsson, Study Director — AstraZeneca R&D, Södertälje, Sweden; Ctril Clarke, MD, Principal Investigator — ICON Development Solutions UK
Locations (1):
- Research Site, Uppsala, Sweden